CLINICAL TRIAL: NCT06882902
Title: Using Forced-response Model and Drift-diffusion Model to Explore OCD's Unique Electroencephalographic Markers of Habit Formation and Expression
Brief Title: Unique Electroencephalography (EEG) Markers of Habit Behaviors in Obsessive-Compulsive Disorder (OCD)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SMHC-OCD-010
Record Dates: First submitted 2024-05-29; First posted 2025-03-19 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: habit; cognitive flexibility; response inhibition
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Habits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Habit formation (Experimental)
  Interventions: Behavioral: habit formation training

INTERVENTIONS:
Behavioral: habit formation training — Participants need to perform habit formation exercises for 4 consecutive days. During the exercises, participants will see a picture stimulus and need to learn the corresponding key press. Each day, participants will spend 30 minutes on the training.

SUMMARY:
This study focuses on explaining the occurrence and development of compulsive behaviors from habit hypothesis. Investigators will study both OCD patients and healthy individuals using Hardwick's forced-response time task(2019), the habit Go/No-Go task, and the Intra-Extra Dimensional Set Shift task. Investigators aim to explore the cognitive abilities and differences between OCD patients and healthy controls in these three tasks. Control variables will include participants' levels of anxiety, depression, and stress, as well as sense of incompleteness and intolerance of uncertainty levels. By examining the differences in habit formation and expression abilities between OCD patients and healthy controls, and exploring the specific brain electroencephalographic activity processes in OCD patients, investigators hope to reveal the abnormal neural activity in habit-related circuits in OCD patients. This could provide new insights for the diagnosis and treatment of OCD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 50;
2. Y-BOCS score greater than or equal to 16;
3. Meet DSM-5 diagnostic criteria with no medication changes in the past two weeks;
4. Right-handed.

Exclusion Criteria:

1. Diagnosed with any DSM-5 disorder other than OCD;
2. Have a major physical illness;
3. Have strong suicidal ideation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of Y-BOCS scores | baseline#after- intervention#1 weeks# (pre-intervention, after intervention, one weeks after intervention)
  We defined the habit training response as the percent reduction of Y-BOCS scores greater than or equal to 35%.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided